CLINICAL TRIAL: NCT00004561
Title: Treatment of Hypertension With Two Exercise Intensities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 129; R01HL056907 (NIH)
Record Dates: First submitted 2000-02-09; First posted 2000-02-10 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
To determine whether exercise training could significantly replace medication as a treatment for mild essential hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Arterial hypertension affects over 50 million Americans. While drug treatment is effective, exercise would be safer, might be cheaper, and would bring added health benefits if it could replace drugs in controlling hypertension.

DESIGN NARRATIVE:

Randomized, controlled trial. Known hypertensives (n=162) whose diastolic blood pressures rose to between 90 and 104 within four months of discontinuing medication under careful observation had their pressures controlled with enalapril. Oxygen consumption (V02) peak was measured during cycle ergometry. Eligible subjects were randomly assigned to 18 months participation in one of three groups: 1) high intensity endurance training (35 minutes three times/week at heart rate at 70-85 percent of V02 peak), 2) moderate intensity endurance training (35 minutes three times/week at heart rate of 50-70 of V02 peak), and 3) contact control. Enalapril was forward or back titrated or discontinued to maintain a normal blood pressure. After 12 months participation, medication was withdrawn under careful supervision from all subjects still taking it. The trial tested the hypotheses that: 1) a greater number of subjects undergoing either or both of the two 18 month exercise training programs would be able to stop anti-hypertensive medication than non-exercising controls, 2) moderate and high intensity endurance training were equally effective in replacing drugs in the treatment of mild essential hypertension, and 3) subjects that were successful at withdrawing anti-hypertensive medication would have: greater improvements in V02 peak, better initial psychological status or greater improvements in psychological status, and greater compliance with the exercise training program.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06; Study Completion 2003-05 (Actual)